CLINICAL TRIAL: NCT03683966
Title: A Structured Survey Among Fabry Patients With a Focus on Adherence to Therapy, Quality of Life and Pain Control
Brief Title: MigALastat Therapy Adherence Among FABRY Patients: A Prospective Multicentral Observational Study
Acronym: MALTA-FABRY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital Muenster (Other); Health Care Center Dr. Markus Cybulla, Muellheim (Unknown)
Responsible Party: Principal Investigator, PD Dr. Peter Nordbeck, Head Consultant Cardiology and Chief of Electrophysiology, Wuerzburg University Hospital
Other Study IDs: AT-IIP-2018
Record Dates: First submitted 2018-09-03; First posted 2018-09-25 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Rare Diseases; Fabry Disease; Adherence, Medication; Quality of Life
Keywords: Fabry; Chaperone therapy; Migalastat; Pharmacological adherence
MeSH Terms: conditions — Rare Diseases; Fabry Disease; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study evaluates adherence to the oral chaperone therapy migalastat in patients with Fabry disease.

DETAILED DESCRIPTION:
Fabry disease is a rare disease and part of the group of lysosomal storage disorders. Since 2016, chaperone therapy as a new therapeutic approach is available.

This study is a prospective cohort study and observes patients under therapy with migalastat. This study is suggested to help estimating the adherence of the oral therapy.

All patients in treatment with migalastat in the Fabry Center Wuerzburg (FAZiT) and selected patients of other cooperating Fabry Centers are included in this study if informed consent is provided.

ELIGIBILITY:
Inclusion Criteria:

* Fabry disease (genetically confirmed)
* Signed informed consent
* 18 years and older

Exclusion Criteria:

* No informed consent
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes every patient with Fabry disease and therapy who is seen in the FAZiT Wuerzburg. Limitation is a therapy with migalastat.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to oral therapy with migalastat according to Medication Assessment Questionnaire | From date of inclusion up to104 weeks (2 years)
  Pharmacological adherence according to adapted and translated 'Medication Assessment Questionnaire'.

SECONDARY OUTCOMES:
Quality of Life according to SF-36 and Wuerzburg pain questionnaire | From date of inclusion up to104 weeks (2 years)
  Change of quality of life under migalastat therapy according to SF-36 and Wuerzburg pain questionnaire. Short Form (36), abbreviated SF-36, is a disease-specific measurement tool for increasing the health-related quality of life. The SF-36 is composed of eight scale-valued domains that correspond to the weighted sums of answers in each section. The range of values of each scale is 0-100 under the assumption that each question has the same weight. A score of 0 is the worst outcome (maximum disability) and a score of 100 is the best outcome (no disability).
  The eight domains of the SF-36 are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.

OTHER OUTCOMES:
Pain according to SF-36 and Wuerzburg pain questionnaire | From date of inclusion up to104 weeks (2 years)
  Change of pain under migalastat therapy according to SF-36 and Wuerzburg pain questionnaire.
  The Wuerzburg pain questionnaire was created by Üçeyler et al. In this questionnaire, the patient's pain phenotype is characterized with questions about the presence of 1) permanent pain, 2) pain attacks, 3) pain crisis, and 4) evoked pain (by touching a cold or warm object or by pressure) in childhood and/or adulthood with the response options Yes, No, or Don't know. Other criteria can be found in the publication (Üçeyler N, Ganendiran S, Kramer D, Sommer C. Characterization of pain in fabry disease. Clin J Pain. 2014 Oct;30(10):915-20.).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nordbeck, MD, PhD, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Wuerzburg University Hospital, Würzburg, Bavaria, Germany

REFERENCES:
- [Background] Muntze J, Salinger T, Gensler D, Wanner C, Nordbeck P. Treatment of hypertrophic cardiomyopathy caused by cardiospecific variants of Fabry disease with chaperone therapy. Eur Heart J. 2018 May 21;39(20):1861-1862. doi: 10.1093/eurheartj/ehy072. No abstract available. PMID 29452394
- [Background] Oder D, Liu D, Hu K, Uceyler N, Salinger T, Muntze J, Lorenz K, Kandolf R, Grone HJ, Sommer C, Ertl G, Wanner C, Nordbeck P. alpha-Galactosidase A Genotype N215S Induces a Specific Cardiac Variant of Fabry Disease. Circ Cardiovasc Genet. 2017 Oct;10(5):e001691. doi: 10.1161/CIRCGENETICS.116.001691. PMID 29018006
- [Background] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102
- [Background] Hughes DA, Nicholls K, Shankar SP, Sunder-Plassmann G, Koeller D, Nedd K, Vockley G, Hamazaki T, Lachmann R, Ohashi T, Olivotto I, Sakai N, Deegan P, Dimmock D, Eyskens F, Germain DP, Goker-Alpan O, Hachulla E, Jovanovic A, Lourenco CM, Narita I, Thomas M, Wilcox WR, Bichet DG, Schiffmann R, Ludington E, Viereck C, Kirk J, Yu J, Johnson F, Boudes P, Benjamin ER, Lockhart DJ, Barlow C, Skuban N, Castelli JP, Barth J, Feldt-Rasmussen U. Oral pharmacological chaperone migalastat compared with enzyme replacement therapy in Fabry disease: 18-month results from the randomised phase III ATTRACT study. J Med Genet. 2017 Apr;54(4):288-296. doi: 10.1136/jmedgenet-2016-104178. Epub 2016 Nov 10. PMID 27834756
- [Background] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681
- [Background] Lenders M, Nordbeck P, Kurschat C, Karabul N, Kaufeld J, Hennermann JB, Patten M, Cybulla M, Muntze J, Uceyler N, Liu D, Das AM, Sommer C, Pogoda C, Reiermann S, Duning T, Gaedeke J, Stumpfe K, Blaschke D, Brand SM, Mann WA, Kampmann C, Muschol N, Canaan-Kuhl S, Brand E. Treatment of Fabry's Disease With Migalastat: Outcome From a Prospective Observational Multicenter Study (FAMOUS). Clin Pharmacol Ther. 2020 Aug;108(2):326-337. doi: 10.1002/cpt.1832. Epub 2020 Apr 27. PMID 32198894
- [Background] Muntze J, Gensler D, Maniuc O, Liu D, Cairns T, Oder D, Hu K, Lorenz K, Frantz S, Wanner C, Nordbeck P. Oral Chaperone Therapy Migalastat for Treating Fabry Disease: Enzymatic Response and Serum Biomarker Changes After 1 Year. Clin Pharmacol Ther. 2019 May;105(5):1224-1233. doi: 10.1002/cpt.1321. Epub 2019 Jan 13. PMID 30506669